CLINICAL TRIAL: NCT01344616
Title: Reducing Preterm Births in Underserved Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PHCC LP (Industry)
Responsible Party: Principal Investigator, James G. Christian, President, PHCC LP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2R44HD047031-02A2 (NIH)
Record Dates: First submitted 2010-07-27; First posted 2011-04-29 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Preterm Birth; Low Birth Weight <2500 Grams; Verylow Birthweight <1500 Grams
Keywords: computer-based behavioral support
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual clinical care (No Intervention): usual clinical care with no intervention
- lifestyle counseling (Experimental): computer-based clinical support to patient
  Interventions: Behavioral: lifestyle support

INTERVENTIONS:
Behavioral: lifestyle support — computer-based lifestyle improvement support and clinician support
  Arms: lifestyle counseling

SUMMARY:
Timely screening and management of modifiable conditions can reduce preterm births, yet providing effective prenatal risk management systems to meet the unique needs of medically underserved populations is complex. If the proposed system proves to be effective in reducing preterm births it can improve maternal and child quality of life as well as reduce the economic burden of preterm births in the U.S.

DETAILED DESCRIPTION:
The primary aim of this proposal is to test the efficacy of a clinic-based, computer-assisted intervention system to significantly reduce preterm births in high-risk populations. This system will: (1) assess a pregnant woman's unique risks in six modifiable areas associated with increased risks of preterm birth including smoking cessation, poor nutrition, domestic violence, maternal depression and stress, urinary and reproductive tract infections and substance use; (2) provide her with tailored advice and action planning tools on reducing her risks; (3) provide her certified nurse midwife or physician with information related to her assessed risks and counseling suggestions tailored for her needs, and [(4) promote effective referrals to, and successful linkages with community-based support organizations.] Because preterm birth rates are much higher for underserved African American women, we are proposing to focus the intervention with this population.

ELIGIBILITY:
Inclusion Criteria: Study inclusion criteria include:

1. age 16-48 years,
2. 1st trimester of pregnancy,
3. race/ethnicity (non-Hispanic Black, or English-speaking Hispanic Black), and 4) a self-reported completion of grade 6 or higher.

Exclusion Criteria: Exclusion criteria include:

1. a medical condition or risk to the pregnancy that the physician or nurse midwife determines serious and a reason for exclusion, and
2. a literacy level of < grade 6. No prior experience using a computer is needed. -

Ages: 16 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 482 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PHCC LP, Pueblo, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Clinical Care | Lifestyle Counseling
Started | 244 | 238
Completed | 209 | 194
Not Completed | 35 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Clinical Care | Lifestyle Counseling | Total
Number analyzed (Participants) | 244 | 238 | 482
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.41 (5.26) | 24.36 (5.18) | 24.4 (5.21)
Sex/Gender, Customized [Number; unit: participants]
  Female | 244 | 238 | 482
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 244 | 238 | 482
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 244 | 238 | 482

OUTCOME MEASURES:

1. Primary Outcome: Birthweight
Description: Birth weight < 2500 grams
Time Frame: 9 months
Population: One Set of twins in the lifestyle counseling arm and 4 sets of twins in the usual clinical care arm
Measure: Number; unit: participants
Arm/Group | Usual Clinical Care | Lifestyle Counseling
Number analyzed (Participants) | 213 | 195
participants | 40 | 26

2. Secondary Outcome: Gestational Weight
Time Frame: 9 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Usual Clinical Care | Lifestyle Counseling
Serious Adverse Events (participants affected / at risk) | 0/244 | 0/233
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No